CLINICAL TRIAL: NCT00960960
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of PI3-Kinase Inhibitor GDC-0941 (Pictilisib) in Combination With Paclitaxel, With and Without Bevacizumab or Trastuzumab, and With Letrozole in Patients With Locally Recurrent Or Metastatic Breast Cancer
Brief Title: A Study of PI3-Kinase Inhibitor GDC-0941 in Combination With Paclitaxel, With and Without Bevacizumab or Trastuzumab, and With Letrozole, in Participants With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDC4629g; GO01304 (Other: Hoffmann-La Roche); 2009-010781-38 (EudraCT Number)
Record Dates: First submitted 2009-08-13; First posted 2009-08-18 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: MBC; PI3K; Avastin; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Letrozole; Paclitaxel; Trastuzumab

ARMS (11):
- Part 1 (Cohort 1-2): Pictilisib 60 mg +Paclitaxel +Bevacizumab (Experimental): Pictilisib 60 mg will be administered orally (PO) once daily (QD) for 21 consecutive days of each 28-day cycle (21+7 schedule) with paclitaxel 90 milligrams per meter square (mg/m^2) intravenously (IV) on Days 1, 8, and 15 and bevacizumab 10 milligrams per kilogram (mg/kg) IV on Days 1 and 15 of each 28-day cycle. In Cohort 1 (Part 1), pictilisib will be evaluated with paclitaxel only; participants in Cohort 1 (Part 1) will be eligible to receive bevacizumab starting at Cycle 2. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Pictilisib; Drug: Paclitaxel
- Part 1 (Cohort 3): Pictilisib 100 mg+ Paclitaxel + Bevacizumab (Experimental): Pictilisib 100 mg will be administered PO QD for 21 consecutive days of each 28-day cycle (21+7 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 and bevacizumab 10 mg/kg IV on Days 1 and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Pictilisib; Drug: Paclitaxel
- Part 2 (Arm A: Cohort 1a): Pictilisib 165 mg + Paclitaxel (Experimental): Pictilisib 165 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity
  Interventions: Drug: Pictilisib; Drug: Paclitaxel
- Part 2 (Arm A: Cohort 2a): Pictilisib 250 mg + Paclitaxel (Experimental): Pictilisib 250 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Pictilisib; Drug: Paclitaxel
- Part 2 (Arm A: Cohort 3a): Pictilisib 330 mg + Paclitaxel (Experimental): Pictilisib 330 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Pictilisib; Drug: Paclitaxel
- Part2(Arm B:Cohort 1b):Pictilisib 200mg+Paclitaxel+Bevacizumab (Experimental): Pictilisib 200 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 and bevacizumab 10 mg/kg IV on Days 1 and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Pictilisib; Drug: Paclitaxel
- Part2(Arm B:Cohort 2b):Pictilisib 250mg+Paclitaxel+Bevacizumab (Experimental): Pictilisib 250 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 and bevacizumab 10 mg/kg IV on Days 1 and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Pictilisib; Drug: Paclitaxel
- Part2(Arm B:Cohort 3b):Pictilisib 260mg+Paclitaxel+Bevacizumab (Experimental): Pictilisib 260 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 and bevacizumab 10 mg/kg IV on Days 1 and 15 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Pictilisib; Drug: Paclitaxel
- Part2(Arm C:Cohort 1c):Pictilisib 180mg+Paclitaxel+Trastuzumab (Experimental): Pictilisib 180 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 and trastuzumab 2-4 mg/kg IV on Days 1, 8, 15, and 22 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Pictilisib; Drug: Paclitaxel; Drug: Trastuzumab
- Part2(Arm C:Cohort 2c):Pictilisib 260mg+Paclitaxel+Trastuzumab (Experimental): Pictilisib 260 mg will be administered PO QD for repeated rounds of 5 consecutive days followed by 2 consecutive drug-free days in each 28-day cycle (5+2 schedule) with paclitaxel 90 mg/m^2 IV on Days 1, 8, and 15 and trastuzumab 2-4 mg/kg IV on Days 1, 8, 15, and 22 of each 28-day cycle. Cycle 1 will be 29 days and subsequent cycles will be 28 days. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Pictilisib; Drug: Paclitaxel; Drug: Trastuzumab
- Part 3: Pictilisib 260 mg + Letrozole (Experimental): Pictilisib 260 mg will be administered PO QD continuously with letrozole 2.5 mg PO QD for each 28-day cycle. Study treatment will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Pictilisib; Drug: Letrozole

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered IV at a dose of 10 mg/kg on Days 1 and 15 of each 28-day cycle.
  Other Names: Avastin
  Arms: Part 1 (Cohort 1-2): Pictilisib 60 mg +Paclitaxel +Bevacizumab; Part 1 (Cohort 3): Pictilisib 100 mg+ Paclitaxel + Bevacizumab; Part2(Arm B:Cohort 1b):Pictilisib 200mg+Paclitaxel+Bevacizumab; Part2(Arm B:Cohort 2b):Pictilisib 250mg+Paclitaxel+Bevacizumab; Part2(Arm B:Cohort 3b):Pictilisib 260mg+Paclitaxel+Bevacizumab
Drug: Pictilisib — Pictilisib will be administered PO QD on escalating doses.
  Other Names: GDC-0941
Drug: Letrozole — Letrozole will be administered PO at a dose of 2.5 mg QD for for each 28-day cycle.
  Arms: Part 3: Pictilisib 260 mg + Letrozole
Drug: Paclitaxel — Paclitaxel will be administered IV at a dose of 90 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle.
  Arms: Part 1 (Cohort 1-2): Pictilisib 60 mg +Paclitaxel +Bevacizumab; Part 1 (Cohort 3): Pictilisib 100 mg+ Paclitaxel + Bevacizumab; Part 2 (Arm A: Cohort 1a): Pictilisib 165 mg + Paclitaxel; Part 2 (Arm A: Cohort 2a): Pictilisib 250 mg + Paclitaxel; Part 2 (Arm A: Cohort 3a): Pictilisib 330 mg + Paclitaxel; Part2(Arm B:Cohort 1b):Pictilisib 200mg+Paclitaxel+Bevacizumab; Part2(Arm B:Cohort 2b):Pictilisib 250mg+Paclitaxel+Bevacizumab; Part2(Arm B:Cohort 3b):Pictilisib 260mg+Paclitaxel+Bevacizumab; Part2(Arm C:Cohort 1c):Pictilisib 180mg+Paclitaxel+Trastuzumab; Part2(Arm C:Cohort 2c):Pictilisib 260mg+Paclitaxel+Trastuzumab
Drug: Trastuzumab — Trastuzumab will be administered IV at a dose of 2-4 mg/kg on on Days 1, 8, 15, and 22 of each 28-day cycle.
  Other Names: Herceptin
  Arms: Part2(Arm C:Cohort 1c):Pictilisib 180mg+Paclitaxel+Trastuzumab; Part2(Arm C:Cohort 2c):Pictilisib 260mg+Paclitaxel+Trastuzumab

SUMMARY:
This is an open-label, multicenter, Phase Ib dose-escalation study to assess the safety, tolerability, and pharmacokinetics of oral (PO) pictilisib administered with letrozole or intravenous (IV) paclitaxel with and without IV bevacizumab or IV trastuzumab in participants with locally recurrent or metastatic breast cancer. The study consists of three parts. Part 1 (pictilisib will be administered in 21+7 schedule along with paclitaxel and/or bevacizumab), Part 2 (pictilisib will be administered in 5+2 schedule along with paclitaxel and/or bevacizumab or trastuzumab) and Part 3 (pictilisib will be administered in combination with letrozole). Part 1 and Part 2 consists of two stages; a dose escalation stage and a cohort-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease
* Adequate organ and bone marrow function as assessed by laboratory tests
* Evaluable disease or disease measurable per RECIST
* Agreement to use an effective form of contraception for the duration of the study

Exclusion Criteria:

* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Any condition requiring full-dose anticoagulants, such as warfarin, heparin, or thrombolytic agents
* Prior anti-cancer therapy (e.g., chemotherapy, biologic therapy, radiotherapy, or hormonal therapy) within 4 weeks or 5 half-lives (whichever is shorter) of the first dose of study treatment
* Uncontrolled current illness
* Active small or large intestine inflammation (such as Crohn's disease or ulcerative colitis)
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
* Known HIV infection
* New York Heart Association (NYHA) Class II or greater congestive heart failure
* Active ventricular arrhythmia requiring medication
* Pregnancy, lactation, or breastfeeding
* Known significant hypersensitivity to study drugs or excipients
* History of arterial thromboembolic disease within 6 months of first study treatment
* No more than two prior chemotherapy regimens for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | First treatment cycle (Day 1 up to Day 29)
Maximum Tolerated Dose (MTD) of Pictilisib | First treatment cycle (Day 1 up to Day 29)
Recommended Phase II Dose (RP2D) of Pictilisib | Baseline up to 54.2 months
Number of Cycles of Each Component of the Treatment Regimen | Baseline up to 54.2 months
Dose Intensity of Each Component of the Treatment Regimen | Baseline up to 54.2 months

SECONDARY OUTCOMES:
Minimum Observed Plasma Concentration (Cmin) of Pictilisib | Parts 1 and 2 (dose escalation): predose (0 hours [h]) on Day (D) 1,3,16, and 17 of Cycle (C) 1. Part 2 (dose expansion): predose (0h) on D3,16,17 of C1; Part 3: Predose (0h) on D1 of C1, C2-6, C≥7, D15 of C1 (cycle length=28 days; up to 54.5 months)
Cmin of Paclitaxel | Parts 1 and 2 (dose escalation): pre-paclitaxel infusion (0 h) on D2 and D16 of C1. Part 2 (dose expansion): pre-paclitaxel infusion (0 h) on D1 and D16 of C1 (cycle length=28 days)
Cmin of Letrozole | Part 3: Predose (0h) on D1 of C1, C2-6, C≥7, D15 of C1 (cycle length=28 days; up to 54.5 months)
Area Under the Curve From Time Zero to Last Measurable Concentrations (AUClast) of Pictilisib | Parts 1 and 2: D1,D3,D16,D17 of C1; study completion. Part 2: D3,D16, D17 of C1; study completion. Part 3: D15 of C1; D1 of C1 to C6, C≥7 (cycle length=28 days; up to 54.5 months) [detailed timeframe is provided in endpoint description]
  Parts 1 and 2 (dose escalation): predose (0 h) and 1,2,3,6 h postdose on D1 and D16 of C1, 24h postdose on D1 of C1; predose (0h) on D3,17 of C1; study completion (up to 55.5 months). Part 2 (dose expansion): predose (0h) and 1,2,3,6h postdose on D16 of C1; predose (0h) on D3, D17 of C1; study completion (up to 55.5 months). Part 3: 3h postdose on D1 of C1; 1,2,3,4,8h postdose on D15 of C1; Predose (0h) on D1 of C1, C2-6, C≥7, D15 of C1 (cycle length=28 days; up to 54.5 months)
AUClast of Paclitaxel | Parts 1 and 2 (dose escalation): D2 and D16 of C1; study completion. Part 2 (dose expansion): D1 and D16 of C1; study completion (cycle length=28 days; up to 55.5 months) [detailed timeframe is provided in endpoint description]
  Parts 1 and 2 (dose escalation): pre-paclitaxel infusion (0 h), end of paclitaxel infusion (infusion length = 60 minutes), end of bevacizumab infusion (infusion length = 30 to 90 minutes), 2,4,6,24 h post-paclitaxel infusion on D2 and D16 of C1; study completion (up to 55.5 months). Part 2 (dose expansion): pre-paclitaxel infusion (0 h), end of paclitaxel infusion (infusion length = 60 minutes), end of bevacizumab infusion (infusion length = 30 to 90 minutes), 1,2,3,6,24 h post-paclitaxel infusion on D1 of C1; pre-paclitaxel infusion (0 h), end of paclitaxel infusion (infusion length = 60 minutes), end of bevacizumab infusion (infusion length = 30 to 90 minutes), 2, 4, 6, 24 h post-paclitaxel infusion on D16 of C1; study completion (cycle length=28 days; up to 55.5 months)
AUClast of Letrozole | Part 3: 1,2,3,4,8h postdose on D15 of C1; Predose (0h) on D1 of C1, C2-6, C≥7, D15 of C1 (cycle length=28 days; up to 54.5 months)
Maximum Observed Plasma Concentration (Cmax) of Pictilisib | Parts 1 and 2: D1,D3,D16,D17 of C1; study completion. Part 2: D3,D16, D17 of C1; study completion. Part 3: D15 of C1; D1 of C1 to C6, C≥7 (cycle length=28 days; up to 54.5 months) [detailed timeframe is provided in endpoint description]
  Parts 1 and 2 (dose escalation): predose (0 h) and 1,2,3,6 h postdose on D1 and D16 of C1, 24h postdose on D1 of C1; predose (0h) on D3,17 of C1; study completion (up to 55.5 months). Part 2 (dose expansion): predose (0h) and 1,2,3,6h postdose on D16 of C1; predose (0h) on D3, D17 of C1; study completion (up to 55.5 months). Part 3: 3h postdose on D1 of C1; 1,2,3,4,8h postdose on D15 of C1; Predose (0h) on D1 of C1, C2-6, C≥7, D15 of C1 (cycle length=28 days; up to 54.5 months)
Cmax of Paclitaxel | Parts 1 and 2 (dose escalation): D2 and D16 of C1; study completion. Part 2 (dose expansion): D1 and D16 of C1; study completion (cycle length=28 days; up to 55.5 months) [detailed timeframe is provided in endpoint description]
  Parts 1 and 2 (dose escalation): pre-paclitaxel infusion (0 h), end of paclitaxel infusion (infusion length = 60 minutes), end of bevacizumab infusion (infusion length = 30 to 90 minutes), 2,4,6,24 h post-paclitaxel infusion on D2 and D16 of C1; study completion (up to 55.5 months). Part 2 (dose expansion): pre-paclitaxel infusion (0 h), end of paclitaxel infusion (infusion length = 60 minutes), end of bevacizumab infusion (infusion length = 30 to 90 minutes), 1,2,3,6,24 h post-paclitaxel infusion on D1 of C1; pre-paclitaxel infusion (0 h), end of paclitaxel infusion (infusion length = 60 minutes), end of bevacizumab infusion (infusion length = 30 to 90 minutes), 2, 4, 6, 24 h post-paclitaxel infusion on D16 of C1; study completion (cycle length=28 days; up to 55.5 months)
Cmax of Letrozole | Part 3: 1,2,3,4,8h postdose on D15 of C1; Predose (0h) on D1 of C1, C2-6, C≥7, D15 of C1 (cycle length=28 days; up to 54.5 months)
Percentage of Participants With Objective Response According to Modified Response Evaluation Criteria in Solid Tumors (RECIST) | Screening up to disease progression or death up to approximately 55.5 months (assessed at Screening and at the end [Days 22-28] of Cycles 2, 5, 8, and 11 and every 3 cycles thereafter [cycle length=28 days; up to approximately 55.5 months])
Duration of Response According to Modified RECIST | Screening up to disease progression or death up to approximately 55.5 months (assessed at Screening and at the end [Days 22-28] of Cycles 2, 5, 8, and 11 and every 3 cycles thereafter [cycle length=28 days; up to approximately 55.5 months])
Percentage of Participants With Death or Disease Progression According to Modified RECIST | Screening up to disease progression or death up to approximately 55.5 months (assessed at Screening and at the end [Days 22-28] of Cycles 2, 5, 8, and 11 and every 3 cycles thereafter [cycle length=28 days; up to approximately 55.5 months])
Progression-free Survival According to Modified RECIST | Screening up to disease progression or death up to approximately 55.5 months (assessed at Screening and at the end [Days 22-28] of Cycles 2, 5, 8, and 11 and every 3 cycles thereafter [cycle length=28 days; up to approximately 55.5 months])

CONTACTS AND LOCATIONS:
Overall Officials: Stina Singel, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (5):
- United States (3):
  - Peoria, Illinois
  - Boston, Massachusetts
  - Nashville, Tennessee
- Leuven, Belgium
- Milan, Lombardy, Italy

REFERENCES:
- [Derived] Schoffski P, Cresta S, Mayer IA, Wildiers H, Damian S, Gendreau S, Rooney I, Morrissey KM, Spoerke JM, Ng VW, Singel SM, Winer E. A phase Ib study of pictilisib (GDC-0941) in combination with paclitaxel, with and without bevacizumab or trastuzumab, and with letrozole in advanced breast cancer. Breast Cancer Res. 2018 Sep 5;20(1):109. doi: 10.1186/s13058-018-1015-x. PMID 30185228